CLINICAL TRIAL: NCT04717713
Title: The Effect of Local Intraoperative Steroid Administration on Post-ACDF Dysphagia - A Prospective Double-Blinded Study by High Resolution Impedance Manometry
Brief Title: The Effect of Local Intraoperative Steroid Administration on Post-ACDF Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202002052MIND
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2021-01

CONDITIONS: Swallowing Function
MeSH Terms: interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- steroid group (Experimental): patients receiving steroid injection for preventing postoperative dysphagia
  Interventions: Drug: steroid injection
- placebo group (Placebo Comparator): patients receiving saline injection for comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: steroid injection — steroid injection at surgical location
  Arms: steroid group
Drug: placebo — saline injection at surgical location
  Arms: placebo group

SUMMARY:
Few methods were available to determine which muscle groups are associated with PD in details in previous investigations. Local steroid administration has shown some effects on PD in a large number meta-analysis. In this study, we aimed to conduct a prospective randomized-double blinded study to exam the efficacy and the safety of the local steroid administration on ACDF patients by using high resolution impedance manometry in patients receiving ACDF.

DETAILED DESCRIPTION:
Postoperative dysphagia (PD) is the most common complication after anterior cervical discectomy and fusion (ACDF). However, few methods were available to determine which muscle groups are associated with PD in details in previous investigations. Local steroid administration has shown some effects on PD in a large number meta-analysis. In this study, we aimed to conduct a prospective randomized-double blinded study to exam the efficacy and the safety of the local steroid administration on ACDF patients, and the also apply the high resolution impedance manometry (HRIM) on patients receiving ACDF for better delineation of the swallowing function. Pressure-flow analysis (PFA), derives pharyngeal pressure flow variables obtained from HRIM were used to analyze the mechanisms of PD.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective anterior cervical spine surgery

Exclusion Criteria:

* patients receiving spine surgery not at the first time
* patients with head and neck cancer
* patients receiving other surgeries at head and neck region
* patients had previous swallowing difficulty history

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
pharyngeal pressure | preoperative, postoperative 1 month
  muscle power at pharyngeal region

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
due to ethic concern